CLINICAL TRIAL: NCT05969002
Title: Pilot Prospective Study for PET-CT Imaging in Participants With Relapsed/Refractory Acute Leukemias
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001620; 001620-C
Record Dates: First submitted 2023-07-31; First posted 2023-08-01 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01-27

CONDITIONS: B Cell; Acute Lymphoblastic Leukemia; Relapsed/Refractory
Keywords: Imaging; Natural History; ACUTE LEUKEMIA
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adult: Participants >/=18 years old with relapsed/refractory B cell ALL proceeding to CAR therapy at the NIH
- Pediatric: Participants <18 proceeding to CAR therapy at the NIH with a clinical indication for FDG PET-CT prior to CAR infusion

SUMMARY:
Background

Acute lymphoblastic leukemia (ALL) accounts for about 25 percent of childhood cancers and for about 20 percent of adult leukemias. The disease can be treated with CAR T-cell infusion but non-central nervous system (CNS) extramedullary disease (EMD) is associated with lower rates of complete remission. 18-fludeoxyglucose (18F-FDG) positron emission tomography-computed tomography (PET-CT) has been shown to be effective for detection of non-CNS EMD in ALL. Pre and post CAR T-cell infusion may help to predict outcomes and risk of early progression.

Objectives

To describe the number of adults with relapsed/refractory B-cell ALL who proceed to CAR T-cell therapy.

Eligibility

Participants >=18 years with relapsed/refractory B-cell ALL who are being screened for CAR T-cell clinical trial enrollment, and

Participants <18 with relapsed/refractory B cell ALL who are being screened for CAR T-cell clinical trial enrollment and have a clinical indication for FDG PET-CT prior to CAR infusion.

Design

Pilot study to add screening FDG PET-CT as part of the pre-CAR T-cell baseline evaluation with additional imaging at day 28 and future timepoints pending evidence of non-CNS EMD on initial scan.

DETAILED DESCRIPTION:
Background

* Acute lymphoblastic leukemia (ALL) is the most common pediatric malignancy, accounting for approximately 25 percent of all childhood cancer. ALL also spans the age spectrum and represents approximately 20 percent of adult leukemias.
* Despite improved survival rates for pediatric, adolescent, and adult ALL, relapse following upfront therapy is common. The recent introduction of chimeric antigen receptor (CAR) T-cell therapies has improved outcomes compared to other available salvage regimens, but limitations to its efficacy exist.
* The presence of non-central nervous system (CNS) extramedullary disease (EMD) at the time of CAR T-cell infusion is associated with lower complete remission (CR) rates compared to isolated medullary disease even with evidence of CAR trafficking to EMD sites. Despite implications for CAR therapy, the true incidence of non-CNS EMD for patients proceeding to CAR is unknown. Our retrospective study estimates the EMD rate to be as high as 21 percent.
* Although 18-fludeoxyglucose (18F-FDG) positron emission tomography-computed tomography (PET-CT) is feasible and has been shown to be high yield for detection of non-CNS EMD in ALL, it is not part of standard evaluation pre-CAR T-cell therapy.
* Recent studies examining the use of pre and post-infusion FDG PET-CT in patients with large cell lymphoma treated with CAR have shown Deauville response criteria, total metabolic tumor volume, and change of standardized uptake values (SUV) to be predictive of CAR T outcomes and risk of early progression. In addition to the use of PET-CT in monitoring CAR T response, circulating tumor DNA (ctDNA) has been shown risk stratify and predict outcomes in large cell lymphoma and can be detected prior to radiographic evidence of relapse.

Objectives

-Describe the proportion of non-CNS EMD in adult participants with relapsed/refractory BALL proceeding to CAR T-cell therapy

Eligibility

* Participants >=18 years with relapsed/refractory B cell ALL who are being screened for CAR T-cell clinical trial enrollment, and
* Participants <18 with relapsed/refractory B cell ALL who are being screened for CAR T-cell clinical trial enrollment and have a clinical indication for FDG PET-CT prior to CAR infusion.

Design

-Pilot study to add screening FDG PET-CT as part of the pre-CAR T-cell baseline evaluation with additional imaging at day 28 and future timepoints pending evidence of non-CNS EMD on initial scan.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Diagnosis: Participants must have a B cell ALL (inclusive of CML with ALL transformation)
* Age: 5-39 years

  * All participants >=18 years old with relapsed/refractory B cell ALL potentially proceeding to CAR therapy at the NIH, or
  * Any participant <18 potentially proceeding to CAR therapy at the NIH with a clinical indication for FDG PET-CT prior to CAR infusion:

    * History of prior EMD
    * History of post-HSCT relapse
    * Clinical signs or incidental findings suspicious for EMD
    * Peripheral disease out of proportion of bone marrow disease burden
* Participants who are breastfeeding or plan to breastfeed must agree to discontinue/postpone breastfeeding within 24 hours of any PET-CT scan
* Ability and willingness of participant or Legally Authorized Representative (LAR) to co-enroll on protocol 10-C-0086 "Comprehensive Omics Analysis of Pediatric Solid Tumors and Establishment of a Repository for Related Biological Studies".
* Ability of participant or Legally Authorized Representative (LAR) to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* Pregnant individuals are excluded from this study
* History of severe, immediate hypersensitivity reaction attributed to compounds of similar chemical or biologic composition to any agents used in study (e.g., FDG injection)

Ages: 5 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2023-08-25 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Proportion of non-CNS EMD in adult participants with relapsed/refractory B-ALL proceeding to CAR T-cell therapy | 3 months
  Estimate the fraction of adult participants who are PET positive for non-CNS EMD

SECONDARY OUTCOMES:
Identify risk factors associated with presence of non-CNS EMD pre-CAR | through 3 months post CAR T
  Risk factors associated with presence of non-CNS EMD
Determine proportion of non-CNS EMD with concurrent CNS disease or history of CNS disease | At time of LP
  Incidence of concurrent CNS disease with non-CNS EMD.

CONTACTS AND LOCATIONS:
Overall Officials: Nirali N Shah, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. In addition, all large scale genomic sequencing will be shared with subscribers to dbGAP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data will be made available during the study and indefinitely. Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Clinical data will be made available upon request and with the permission of the study PI. Genomic data are made available via dbGAP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_001620-C.html